CLINICAL TRIAL: NCT04916093
Title: Safety and Efficacy of Sitagliptin, Vildagliptin, and Metformin in Recently Diagnosed Drug-naïve Patients With Type 2 Diabetes
Brief Title: Safety and Efficacy of Antidiabetic Drugs in Recently Diagnosed Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Beni-Suef University (Other)
Collaborators: Minia University (Other)
Responsible Party: Principal Investigator, Asmaa Abdelfattah Elsayed, PHD candidate in clinical pharmacy department and PI, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MinyaU
Record Dates: First submitted 2021-05-24; First posted 2021-06-07 (Actual); Last update posted 2021-06-07 (Actual); Status verified 2021-06

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Vildagliptin; Sitagliptin Phosphate; Metformin; Tablets

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Sitagliptin Group (Experimental): Included 20 recently diagnosed type 2 diabetic subjects. They all received sitagliptin 100 mg therapy once daily before breakfast.
  Interventions: Drug: Sitagliptin 100mg
- Vildagliptin Group (Experimental): Included 20 recently diagnosed type 2 diabetic subjects. They all received vildagliptin 50 mg therapy twice daily before breakfast and supper.
  Interventions: Drug: Vildagliptin 50 MG
- Metformin Group (Active Comparator): Included 20 recently diagnosed type 2 diabetic subjects. They all received control 1 gm twice daily
  Interventions: Drug: MetFORMIN 1000 Mg Oral Tablet

INTERVENTIONS:
Drug: Vildagliptin 50 MG — Galvus 50 mg oral tablets
  Arms: Vildagliptin Group
Drug: Sitagliptin 100mg — Januvia 100mg oral tablets
  Arms: Sitagliptin Group
Drug: MetFORMIN 1000 Mg Oral Tablet — Glucophage 1000 mg oral tablets
  Arms: Metformin Group

SUMMARY:
The current study aims to investigate Sitagliptin and vildagliptin efficacy and safety compared to metformin as 1st line options for T2D patients.

DETAILED DESCRIPTION:
This is a randomized case-controlled study in which drug-naive type-2 diabetic patients were divided into 3 groups and followed up for three months.

ELIGIBILITY:
Inclusion Criteria:

* Recently diagnosed type2 diabetic adult subjects who were not on an oral hypoglycemic drug (OHA) at the screening visit were eligible to participate.

Exclusion Criteria:

1. Type1 diabetes or ketoacidosis
2. End-organ failure as chronic renal failure (estimated serum creatinine level ≥ 1.5mg/dl in male and ≥ 1.4mg/dl in female)
3. Liver cell failure (elevated alanine transaminase (ALT ) and/or aspartate transaminase (AST) ≥ 2 folds)
4. Any stage of heart failure
5. Previous history of pancreatitis
6. Previous history of taking medication which may alter the efficacy of either drug eg: (other OHA drug, corticosteroids, and oral contraceptives)
7. Pregnant or lactating females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 60 (Actual)
Dates: Start 2019-12-20 (Actual); Primary Completion 2020-06-10 (Actual); Study Completion 2020-12-15 (Actual)

PRIMARY OUTCOMES:
Changes in glycemic parameters | 3-months
  serum fasting glucose (mg/dl), and 2-hr postprandial glucose (mg/dl)
Changes in Serum insulin (IU/l) | 3-months
  using enzyme immunoassay (EIA) kits
Insulin resistance | 3-months
  measured by HOMA model assessment (HOMA-IR) using the following formula: (Fasting insulin (IU/ml) × Fasting glucose (mg/dl))/405
Beta cell function (HOMA-B) | 3-months
  measured by (360 ×Fasting Insulin (IU/ ml) )/(Fasting glucose(mg/dl)-63)
Changes in HbA1c (%) | 3-months
  Changes in HbA1c (%)

SECONDARY OUTCOMES:
Changes in Lipid profile | 3-months
  (total cholesterol, TG, HDL, and LDL) (mg/dl)
Changes in liver enzymes | 3-months
  ALT and AST (U/l)
Changes in Renal function tests | 3-months
  creatinine and urea (mg/dl)

CONTACTS AND LOCATIONS:
Overall Officials: Asmaa A Elsayed, Master, Principal Investigator — BUC
Locations (1):
- Minya University Hospital, Minya, Egypt

IPD SHARING:
Plan to Share IPD: No